CLINICAL TRIAL: NCT04669314
Title: Surgical Approach in Liver Hemangiomas With Special Emphasis on Lesion Diameter and Type of Surgery
Brief Title: Surgical Approach in Liver Hemangiomas
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Elvan Onur Kirimker, M.D., Ankara University
Other Study IDs: AUTF-Hemangioma
Record Dates: First submitted 2020-12-02; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Hemangioma Liver
Keywords: hemangioma; liver resection; enucleation
MeSH Terms: conditions — Hemangioma | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Liver resection or enucleation for liver hemangioma — Operations in which the hemangioma is selectively removed from the liver parenchyma border are named enucleation, and the operations in which the hemangioma is removed anatomically or non-anatomically with some liver parenchyma surrounding it are named liver resection

SUMMARY:
Operations performed for liver hemangioma between January 2017 and December 2018 will be retrospectively analyzed.

DETAILED DESCRIPTION:
Operations performed for liver hemangioma at Ankara University Hospitals will be retrospectively analyzed. Patient and disease characteristics including demographics, laboratory tests, imaging studies, type of surgical approach and outcomes including postoperative laboratory tests, record of complications, duration of hospital stay will be reviewed. Complications were classified according to Clavien-Dindo classification. The patients were informed about the surgeries in advance and their informed consents about surgeries and data collection for scientific purposes were obtained. Datafile will be anonymized before analysis and original file will be destroyed. Outcomes such as complications, hospital stay, blood transfusion and mortality will be compared between groups created according to type of surgery, lesion size, preoperative laboratory values and demographic features. Variables for prediction of better outcomes are expected to be discovered.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent surgery for liver hemangioma

Exclusion Criteria:

* Cases lacking of more than 20% of critical data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients underwent surgery for liver hemangioma between 2007 and 2018 at Ankara University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Complications | Complications reported within 3 months after surgery will be evaluated within 15 days after completion of data collection
  Complications after surgery for hemangioma will be collected from records and and will be classified according to 'The Clavien-Dindo Classification of Surgical Complications'. The classification grades are ranging between Grade 1(better) which indicates minor deviation from normal postoperative course and Grade 5 (worst) which means death as a complication.

SECONDARY OUTCOMES:
Hospital stay | Hospital stay starting with operation and ends with discharge will be compared within 15 days after completion of data collection
  Length of hospital stay postoperatively
Transfusion | Erythrocyte transfusion during surgery will be analyzed within 15 days after completion of data collection
  Rate of erythrocyte transfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Ibni Sina Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Study protocol will be seen on clicaltrials.gov